CLINICAL TRIAL: NCT02377531
Title: Gestational Diabetes Mellitus: Does Early Screening and Treatment for Patients at Increased Risk for Gestational Diabetes Impact Perinatal Outcomes? A Randomized Controlled Trial
Brief Title: Early Screen and Treatment for Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00020026
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes
Keywords: early glucose screen, perinatal outcome
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early glucose screen group (Other): Participants with high risk factors for gestational diabetes, will be randomly assigned to an early glucose screen group: it consists of an oral load of 50 grams of glucose followed by a measurement of serum glucose 1 hour later, and if abnormal (higher than 130mg/dl), will undergo a 100 gram oral load of glucose followed by serum glucose levels drawn 1,2 and 3 hours after the load. If abnormal according to Carpenter-Cousant criteria, the participant will undergo standard of care for Gestational Diabetes.
  Interventions: Other: Early glucose screen group
- Standard glucose screen group (Other): The participants in this group will be randomized to undergo the testing process previously described at 24 to 28 weeks.
  Interventions: Other: Standard glucose screen group

INTERVENTIONS:
Other: Early glucose screen group — Main intervention is randomization: half of the participants will be randomized to undergo a 50 gram oral glucose load with a 1 hour serum glucose measurement as a screen for Gestational Diabetes mellitus at 12 to 18 weeks of pregnancy instead of standard 24 to 28 weeks of pregnancy
  Arms: Early glucose screen group
Other: Standard glucose screen group — Main intervention is randomization: half of the participants will be randomized to undergo a 50 gram oral glucose load with a 1 hour serum glucose measurement as a screen for Gestational Diabetes mellitus at 24 to 28 weeks of pregnancy
  Arms: Standard glucose screen group

SUMMARY:
In the current study we aim to determine if early glucose screening and treatment among women at high risk for GDM improves perinatal outcome and decreases gestational weight gain. Half of the participant will be assigned to an early glucose screen group (12-18 weeks) and treatment if necessary and the other half to a standard 24-28 weeks glucose screen.

ELIGIBILITY:
Inclusion Criteria:

Pregnant subjects 18-45 y/o and Any of the following:

Obesity defined as having a BMI>30 kg/m2 History of pregnancy complicated with GDM History of pregnancy complicated with macrosomia First degree relative with diabetes Multiple gestation

Exclusion Criteria:

* Incomplete Data: if any data is missing (i.e Delivery data) , analysis cannot be completed.

Pregnancy complicated with fetal malformations or aneuploidy: It affects prenatal care, mode of delivery as well as perinatal outcome.

Pregestational or Overt Diabetes: Patients with Diabetes cannot be diagnosed with GDM.

Chronic medical conditions such as hypertension, renal disease, autoimmune conditions: Those conditions may affect prenatal care, perinatal morbidity.

Early diabetes screen performed prior to enrollment in study: Participant cannot be randomized, and probably have been treated.

Medical contraindication to glucose tolerance test (bariatric surgery): patients with h/o gastric bypass frequently cannot tolerate oral glucose load, therefore cannot be screened for GDM in the traditional way.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1020 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Composite Perinatal morbidity | up to 28 days after birth
  The primary study outcome is a composite of perinatal morbidities including perinatal mortality (stillbirth or neonatal death), neonatal hypoglycemia, hyperbilirubinemia, and birth trauma. Transcutaneous bilirubin is routinely measured at Tampa General Hospital (TGH) on all babies at least once. A value greater than the 95th percentile for or need for phototherapy at any given point after birth will be considered an elevated level. Birth trauma is defined as brachial plexus palsy or clavicular, humeral, or skull fracture.

SECONDARY OUTCOMES:
Maternal weight gain | up to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rodriguez, MD, Principal Investigator — University of South Florida; Judette Louis, MD, MPH, Study Chair — University of South Florida; Linda Odibo, Study Director — University of South Florida
Locations (2):
- United States (2):
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - TGH Health Park Genesis Clinic, Tampa, Florida